CLINICAL TRIAL: NCT00208923
Title: Allogeneic Bone Marrow Transplantation With Matched Unrelated Donors for Patients With Hematologic Malignancies Using a Preparative Regimen of Busulfan, Cyclophosphamide, and Fludarabine
Brief Title: Allogeneic Bone Marrow Transplantation With Matched Unrelated Donors for Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Amelia A Langston, MD, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0709-1997
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Hematologic Malignancies
Keywords: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Busulfan; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Chemotherapy-only conditioning regimen comprising busulfan (Bu), cyclophosphamide (Cy) and fludarabine (FLUDARA) followed by an allogeneic stem cell transplant.
  Interventions: Drug: Busulfan, Cyclophosphamide and Fludarabine

INTERVENTIONS:
Drug: Busulfan, Cyclophosphamide and Fludarabine — * Bulsufan 1mg/kg/dose P.O. every 6 hours for 4 days. If intravenous, busulfan dose will be 0.8 mg/kg every 6 hours for 16 doses.
  * Fludarabine 40 mg/m2 a day for 5 days via IV over 2 hours, dose based on weight.
  * Cyclophosphamide given via IV over 1 hour at dose of 60 mg/kg/day for 2 consecutive days.

SUMMARY:
Patients who have cancer of the bone marrow (leukemia) or lymph gland (lymphomas) are being asked to take part in this study. This study uses a new chemotherapy regimen and matched volunteer stem cell transplant to treat patients with cancers of this kind.

DETAILED DESCRIPTION:
Patients who have cancer of the bone marrow (leukemia) or lymph gland (lymphomas) are being asked to take part in this study. This study uses a new chemotherapy regimen and matched volunteer stem cell transplant to treat patients with cancers of this kind.

High dose chemotherapy, followed by a transplant of stem cells collected from either bone marrow (BMT) or peripheral blood of an HLA (tissue type) matched unrelated donor, offers a potential cure for several serious blood diseases including acute and chronic leukemia, myelodysplastic syndrome and lymphoma.

However, the success of allogeneic (unrelated volunteer matched donor) transplant is limited by treatment related illness, death, and relapse in patients with refractory (resistant) disease and/or advanced age (older than 40 years).

Patients being sought for this study do not have an HLA-matched relative to donate stem cell; however, through The National Marrow Donor Program or International Registries, an HLA-matched unrelated donor has been found to donate stem cells. Preliminary data shows that the outcome is comparable between bone marrow and peripheral blood stem cell transplantations, and donor preference will determine which type of cells the patient receives.

To carry out an unrelated transplant, a normal person with similar HLA type must be available to donate cells. The patient must be prepared to accept the donor cells by decreasing the body's immune systems. In addition, the malignant (cancerous) cells must be destroyed to allow growth and repopulation of healthy donor cells. This is usually done by giving total body irradiation and chemotherapy, which is associated with severe side effects in patients over age 40.

In other studies, it has been found that treating the patient with two anticancer drugs, Busulfan and Cyclophosphamide, without total body irradiation, is safe and sufficiently immunosuppressive. High dose Busulfan and Cyclophosphamide are frequently used in combination prior to matched related bone marrow transplant in case of acute leukemia, myelodysplastic syndrome (MDS), Hodgkin's disease (HD), and chronic myeloid leukemia (CML). Fludarabine (another anticancer drug) suppresses the immune system and has strong anticancer effect against chronic lymphocytic leukemia (CLL) and non-Hodgkin's lymphoma (NHL). Researchers are studying a new chemotherapy regimen that includes fludarabine, along with busulfan and cyclophosphamide, to provide more immunosuppression and anti-cancer effect without increasing the chemotherapy related toxicity in patients with CML, acute leukemia and MDS, CLL, NHL, and HD.

The purposes of this study are: 1) to decrease the side effects due to the chemotherapy used to treat the bone marrow; and 2) to increase the number of tumor cells killed. There will be up to 55 patients enrolled in this study at Emory University. The expected duration of each subject's participation in this study will be for two years.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to participate in this study must have CML in the first chronic phase, AML in the first complete remission, AML in second remission, ALL or hybrid leukemia in the first complete remission, ALL in second remission, or advanced MDS. Final eligibility for this study will be determined by the health professionals conducting the trial.

Exclusion Criteria:

* Patients with active CNS malignant disease, or an invasive/systemic fungal infection are not eligible to participate in this study. Patients who are lactating, or who have an HLA identical or 1 antigen mismatched relative who is eligible and willing to donate bone marrow will also be excluded from the study. Final eligibility for this study will be determined by the health professionals conducting the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 1998-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Assess activity of preparative regimen in patients with CML, AML, RAEB, RAEB-t, CLL, NHL, HD, in all patients with refractory anemia, ringed sideroblasts, undergoing allogeneic stem cell transplantation from volunteer matched unrelated donor (VUD). | 6 months

SECONDARY OUTCOMES:
Determine disease-free and overall survival. | 2 years+

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Langston, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory Universtiy Winship Cancer Institute, Atlanta, Georgia, United States